CLINICAL TRIAL: NCT04060771
Title: Prospective, Double-blind Study Comparing Palonosetron and Dexamethasone in the Prophylaxis of Post-Operative Nausea and Vomiting in Children Submitted to Strabismus Surgery
Brief Title: Post-Operative Nausea and Vomiting in Children Submitted to Strabismus Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Alexandra Rezende Assad, PhD, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Strabismus surgery
Record Dates: First submitted 2019-04-18; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia; Strabismus; PONV
Keywords: Anesthesia; Strabismus; PONV
MeSH Terms: conditions — Strabismus; Postoperative Nausea and Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be divided between two groups, Group P will receive single dose of palonosetron whereas Group D will receive a single dose of dexamethasone during general anesthesia.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Experimental): During general anesthesia patients will receive a single intravenous dose of palonosetron 1 mcg.Kg-1.
  Interventions: Drug: Palonosetron
- Group D (Active Comparator): During general anesthesia patients will receive a single intravenous dose of dexamethasone 0.2 mg.Kg-1.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Palonosetron — prophylaxis of postoperative nausea and vomiting
  Other Names: Prophylactic
  Arms: Group P
Drug: Dexamethasone — prophylaxis of postoperative nausea and vomiting
  Other Names: Prophylactic
  Arms: Group D

SUMMARY:
Background: Postoperative nausea and vomiting (PONV) is one of the main causes of patient and family dissatisfaction, which may delay the onset of oral intake and postpone discharge. In pediatric patients, the incidence of PONV is high, and in some studies it can reach values of 70%. Strabismus surgery is considered an independent risk factor for PONV. Palonosetron is a second generation antiemetic drug, 5-hydroxytryptamine receptor antagonist, with a long half-life, which allows single dose administration and has been shown to be safe and effective in the treatment of chemotherapy induced nausea and vomiting, and has been used with satisfactory results in the prophylaxis of PONV in adult and pediatric patients. Studies involving palonosetron are still scarce.

DETAILED DESCRIPTION:
Prospective, double-blind study comparing Palonosetron and Dexamethasone in the prophylaxis of Post-Operative Nausea and Vomiting in children submitted to Strabismus surgery ABSTRACT Background: Postoperative nausea and vomiting (PONV) is one of the main causes of patient and family dissatisfaction, which may delay the onset of oral intake and postpone discharge. In pediatric patients, the incidence of PONV is high, and in some studies it can reach values of 70%. Strabismus surgery is considered an independent risk factor for PONV. Palonosetron is a second generation antiemetic drug, 5-hydroxytryptamine receptor antagonist, with a long half-life, which allows single dose administration and has been shown to be safe and effective in the treatment of chemotherapy induced nausea and vomiting, and has been used with satisfactory results in the prophylaxis of PONV in adult and pediatric patients. Studies involving palonosetron are still scarce.

Objective: The study aims to compare the incidence of PONV after intravenous administration of palonosetron or dexamethasone in pediatric patients undergoing elective strabismus surgery under general anesthesia.

Materials and Methods: This prospective, double-blind study consist of 80 patients of both genders, classified as ASA grade I and II, ranging in age from 2 to 15 years, scheduled for elective strabismus surgery at Hospital Universitário Antonio Pedro(HUAP), after consent by their parents. Patients will be randomized into two groups of 40 patients each. Group P will receive intravenous dose of palonosetron (1 mg.kg-1), and Group D will receive dexamethasone (0.2 mg.kg-1) after induction of anesthesia. Pacients will be observed for 6 hours before discharge and post-discharge symptoms will be assessed through telephone survey after 24 and 48 hours. At the end of the study, results will be compiled and statistical analysis will be done by using Mann-Whitney test, Chi-squared test and Fisher test.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing elective strabismus surgery
* Physical state according to an American Society of Anesthesiologists (ASA) I and II

Exclusion Criteria:

* Children nor involved in surgery
* Participation in another study in the last month
* Previous history of PONV
* Occurrence of episodes of nausea or vomiting in the last 24 hours before surgery
* Chronic use of corticosteroids
* Previous history of motion sickness
* Use of psychoactive drugs or any other medicine with an antiemetic effect;
* Known hypersensitivity to any study medication
* Severe diseases in organs such as kidney, liver, lung, heart, brain and bone marrow

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Vomiting | 48 hours postoperative
  Quantify the frequency of individual episodes of vomiting at the first 48 hours after surgery.

SECONDARY OUTCOMES:
Vomiting | 24 hours postoperative
  Quantify the frequency of individual episodes of vomiting at the first 24 hours after surgery.
Vomiting | 6 hours postoperative
  Quantify the frequency of individual episodes of vomiting at the first 6 hours after surgery.
Vomiting | 2 hours postoperative
  Quantify the frequency of individual episodes of vomiting at the first 2 hours after surgery.
Nausea | 48 hours postoperative
  Quantify the frequency of episodes of nausea at the first 48 hours after surgery.
Nausea | 24h hours postoperative
  Quantify the frequency of episodes of nausea at the first 24 hours after surgery.
Nausea | 6h hours postoperative
  Quantify the frequency of episodes of nausea at the first 6 hours after surgery.
Nausea | 2h hours postoperative
  Quantify the frequency of episodes of nausea at the first 2 hours after surgery.
Check adverse effects | 48 hours postoperative
  Check the frequency of adverse events (headache, dizziness, drowsiness).
Treatment cost | 48 hours postoperative
  Price evaluation of antiemetic drugs.
Response to medication | 48 hours postoperative
  Quantify the number of complete responders (individuals who did not have an episode of PONV and did not require rescue medication).

CONTACTS AND LOCATIONS:
Overall Officials: Júlio CA Moreira, MD, Principal Investigator — Hospital Universitário Antonio Pedro
Locations (1):
- Hospital Universitário Antonio Pedro, Niterói, Rio de Janeiro, Brazil